CLINICAL TRIAL: NCT06809036
Title: Mobilisation and Breathing Exercises After Abdominal Surgery at Sahlgrenska University Hospital
Acronym: SUMO
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: FoU i VGR no: 284167
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard practice: Routine of postoperative mobilisation and breathing exercises will recorded
- Optimised practice: Postoperative mobilisation and breathing exercises will be recorded after a co-creation process where optimal practice is defined and implemented

SUMMARY:
The aim of the study is to evaluate the effect of a new care strategy, including earlier and more intensive mobilization and individually adapted breathing exercises, regarding length of stay, recovery, complications and which factors predict interventions early in the postoperative course after various abdominal surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective or emergency open, or robot-assisted abdominal surgery
* has an expected anesthesia time of over 4 hours
* is extubated on the operating table
* planned overnight stay in the postoperative ward.

Exclusion Criteria:

* plastic, trauma, transplant or orthopedic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Sahlgrenska university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time in postoperative care | At discharge from postoperative care up to two days after surgery.
  Actual time from arrival to, to discharche from postoperative care.

SECONDARY OUTCOMES:
Time to first mobilisation | Up to the second postoperative day
  Time from arrival to postoperative care to first mobilisation
Time to start of breathing exercises | Up to the second postoperative day
  Time from arrival to postoperative care until start of specific breathing exercises.

OTHER OUTCOMES:
Number of mobilisations | Up to the second postoperative day
  Number of mobilisations
Number of sessions of breathing exercises | Up to the second postoperative day
  Number of sessions of breathing exercises
Time at hospital | At discharge from the hospital up to four weeks after surgery
  Time from the day of surgery to discharge from hospital.
Type of mobilisation | Up to the second postoperative day
  Registration of type of mobilisation
Type of breathing exercises | Up to the second postoperative day
  Type of breathing exercises prescribed
Analgesia | Up to the second postoperative day
  Type of analgesia
Complications | At discharge from the hospital up to four weeks after surgery.
  Postoperative pulmonary complications.
Dose of analgesia | Up to the second postoperative day
  Dose of analgesia given

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
It is not included in the ethical approvement